CLINICAL TRIAL: NCT00999414
Title: Compassionate Use Study of Carfilzomib for Patients With Relapsing or Resistant Multiple Myeloma
Brief Title: UARK 2009-32 Compassionate Use Study of Carfilzomib
Acronym: 2009-32
Status: No longer available | Type: Expanded Access
Sponsor: University of Arkansas (Other)
Collaborators: Onyx Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 111527
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Multiple Myeloma
Keywords: MM
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib (20mg/m2) IV push to be given at maximum rate of 10ml/minute on Days 1 and Day 2 of Cycle 1 only.
  Carfilzomib (27mg/m2) IV bolus to be given at maximum rate of 10ml/minute on Day 8, 9, 15, and 16 of Cycle 1, then through Cycle 2 and beyond if initial dosing with 20mg/m2 tolerated.
  For patients who tolerated 27mg/m2 through cycle 2 Days 1 and 2, Carfilzomib dose may be escalated to 36mg/m2 on days 8, 9, 15 and 16 of cycle 2. If tolerated, subsequent cycles will utilize 36mg/m2.

SUMMARY:
This is a compassionate use, open-label, IND study for the purpose of providing carfilzomib to patients with relapsed or resistant refractory multiple myeloma.

DETAILED DESCRIPTION:
The protocol has been designed for relapsing or refractory multiple myeloma patients. A maximum of 30 patients may be treated on this protocol.

Since this is a compassionate use study of an investigational agent, the size is determined by agreement with the manufacturer of carfilzomib. Therefore, the time period for enrollment and accrual number will be limited to N=30.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically documented multiple myeloma which is relapsing or resistant after stem cell transplantation, or when other conventional therapies have failed or are contraindicated
* Serum creatinine < 3.0 mg/dL OR calculated creatinine clearance >15 mL/min calculated or measured clearance is ≥15 mL/min
* ANC > 1000/mm3 (may be supported with growth factors)
* Platelet count > 30,000/mm3 (may receive transfusion)
* Female participant of child-bearing potential has agreed to use dual methods of contraception for the duration of the study
* Male participant has agreed to use a barrier method of contraception if sexually active with a female of child-bearing potential
* Patients must have signed and IRB-approved written informed consent form and demonstrate willingness to meet follow-up schedule and study procedure obligations

Exclusion Criteria:

* Active infection requiring systemic treatment
* Requires concomitant use of approved or investigative anticancer therapeutic treatment with activity against multiple myeloma, other than dexamethasone
* Concomitant use of other investigative agents (e.g., antibiotics or antiemetics)
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2009-11; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Barlogie, MD, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- See also: MIRT Clinical Trials — http://www.myeloma.uams.edu/